CLINICAL TRIAL: NCT01205789
Title: EXCEL Clinical Trial (Universal Registry)
Acronym: EXCEL
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-389 UR
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Coronary Occlusion; Left Main Coronary Artery Disease; Stent Thrombosis; Vascular Disease; Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: Drug eluting stents; Stents; Angioplasty; Left Main Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Restenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Universal Registry: Subjects who are either not eligible for randomization or for other reasons are not randomized will be consented for the Universal Registry

SUMMARY:
The purpose of the Universal Registry is to assess the proportion and reasons for which subjects with angiographically significant ULMCA disease requiring revascularization during the time course of this study are not randomized; to compare the baseline characteristics of subjects; and to assess the variability in randomization eligibility and treatment patterns.

DETAILED DESCRIPTION:
Approximately 100 consecutive subjects who otherwise meet all enrollment criteria, will be analyzed separately as intermediate lesion subjects, and will be followed through the time of initial treatment per standard of care with intended PCI, CABG or medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are either not eligible for randomization or for other reasons are not randomized will be consented for the Universal Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1000 consecutive subjects enrolled which includes approximately 100 consecutive subjects with intermediate lesions
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
This study has no Primary outcome measure, it is an observational study to collect information on subjects not randomized to the RCT portion of the study. | At the time of enrollment into the study
  The purpose of the Universal Registry is to assess the proportion and reasons for which subjects with angiographically significant ULMCA disease requiring revascularization during the time course of this study are not randomized; to compare the baseline characteristics of subjects; and to assess the variability in randomization eligibility and treatment patterns.
  There are no follow-up time points for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W Stone, MD, Principal Investigator — Columbia University; Patrick W Serruys, MD, Principal Investigator — Erasmus Medical Center; Joseph Sabik, MD, Principal Investigator — Cleveland Clinical Main Campus; A. Pieter Kappetein, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Abbott Vascular, Santa Clara, California, United States